CLINICAL TRIAL: NCT02084199
Title: Study to Evaluate the Pharmacokinetics, Safety, Tolerability of 100 mg Multiple Doses of GLPG0634 in Subjects With Renal Impairment Compared to Healthy Subjects
Brief Title: Study to Evaluate GLPG0634 in Subjects With Renal Impairment Compared to Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GLPG0634-CL-106; 2013-004407-40 (EudraCT Number)
Record Dates: First submitted 2014-03-09; First posted 2014-03-11 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Part 1 - Severe renal impairment (Experimental): Part 1 - Group 1: subjects with severe renal impairment or end-stage renal disease (ESRD), not on dialysis: Estimated glomerular filtration rate (eGFR) between 15-29 mL/min/1.73 m2 or <15 mL/min/1.73m² will be administered GLPG0634 100 mg once daily for 10 days
  Interventions: Drug: GLPG0634
- Part 1: Normal renal function (Experimental): Part 1 - Group 2: subjects with normal renal function: eGFR ≥90 mL/min/1.73m² will be administered GLPG0634 100 mg once daily for 10 days
  Interventions: Drug: GLPG0634
- Part 2 - Mild renal impairment (Experimental): Part 2 - Group 3: subjects with mild renal impairment: eGFR between 60-89 mL/min/1.73 m² will be administered GLPG0634 100 mg once daily for 10 days
  Interventions: Drug: GLPG0634
- Part 2 - Moderate renal impairment (Experimental): Part 2 - Group 4:subjects with moderate renal impairment: eGFR between 30-59 mL/min/1.73 m² will be administered GLPG0634 100 mg once daily for 10 days
  Interventions: Drug: GLPG0634
- Part 2 - Normal renal function (Experimental): Part 2 - Group 5: subjects with normal renal function: eGFR ≥90 mL/min/1.73 m² will be administered GLPG0634 100 mg once daily for 10 days
  Interventions: Drug: GLPG0634

INTERVENTIONS:
Drug: GLPG0634 — 100 mg oral tablet, intake once daily for 10 days
  Other Names: GLPG0634 tablets

SUMMARY:
This will be an open label study to assess the influence of renal impairment on the pharmacokinetics (PK) of GLPG0634 and its metabolite after once daily oral administrations of 100 mg GLPG0634 for 10 days in subjects with renal impairment and matched healthy controls.

Also, safety and tolerability of once daily oral doses of GLPG0634 for 10 days in subjects with renal impairment and matched healthy controls will be evaluated.

DETAILED DESCRIPTION:
The study will be divided in two parts.

In Part 1, 3 subjects with severe renal impairment or end-stage renal disease (ESRD) not yet requiring dialysis (Group 1) will be recruited first. Thereafter, 3 subjects with normal renal function (Group 2) will be recruited. If a substantial effect on the PK in renal impaired subjects is observed on Day 10, the sponsor may elect to stop Part 1 of the study without enrolling the complete set of subjects and Part 2 will be initiated. In case no substantial effect on the PK is observed, 3 further subjects in both Group 1 and 2 will be recruited and analysed. If a substantial effect on the PK is observed, the study will proceed to Part 2. Part 2 of the study will not be conducted, if in Part 1 no substantial difference in PK is seen.

In Part 2, Group 3 (mild renal impairment) and Group 4 (moderate renal impairment) will be recruited first. After completion of the mild and moderate impairment groups, Group 5 (normal renal function) will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Male and female white subjects between 18-79 years of age (inclusive)
* Subjects must have a BMI between 18-34 kg/m², inclusive
* Part 1, Group 1: subject with severe renal impairment or ESRD, not on dialysis : eGFR between 15-29 mL/min/1.73 m2 or <15 mL/min/1.73m²
* Part 1, Group 2: subject with normal renal function: eGFR ≥90 mL/min/1.73m²
* Part 2, Group 3: subject with mild renal impairment: eGFR between 60-89 mL/min/1.73 m²
* Part 2, Group 4:subject with moderate renal impairment: eGFR between 30-59 mL/min/1.73 m²
* Part 2, Group 5: subject with normal renal function: eGFR ≥90 mL/min/1.73 m²
* Subjects must be judged to be in good health (subjects with normal renal function)/in a stable condition and acceptable for study participation (subjects with renal impairment) based upon the results of a medical history, physical examination, vital signs, 12-lead ECG, and laboratory profile

Exclusion Criteria:

* A subject with a known hypersensitivity to ingredients of the study medication or a significant allergic reaction to any drug
* Subject has previously participated in a GLPG0634 study or has previously received GLPG0634
* Concurrent participation or participation within 8 weeks prior to the initial study drug administration in a drug/device or biologic investigational research study
* A subject with active drug or alcohol abuse within 2 years prior to the initial study drug administration
* A subject who has a current child wish
* Female subject less than 6 months post-partum, post-abortion or post-lactation prior to study drug administration or is pregnant or breastfeeding

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  Cmax of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Area under the plasma drug concentration-time curve over 24 hours (AUC0-24h) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  AUC0-24h of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function

SECONDARY OUTCOMES:
Cumulative amount excreted in urine expressed in μg and % of the dose administered (Ae) | Between dosing on Day 1 up to 48 h after dosing on Day 10 (Day 12)
  Ae of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Renal clearance (CLR) | Between dosing on Day 1 up to 48 h after dosing on Day 10 (Day 12)
  CLR (calculated as Ae/AUC, where Ae and AUC are calculated over the same interval) of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Plasma concentration observed at 24 h post-dose (C24h) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  C24h of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Average plasma concentration (Cavg) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  Cavg (calculated as AUC0-24h/24h) of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Time of occurrence of Cmax (tmax) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  Tmax of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Area under the plasma drug concentration-time curve from zero to the last sampling time at which concentrations were at or above the limit of quantification (AUC0-z) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  AUC0-z of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Area under the plasma drug concentration-time curve, extrapolated to infinity (AUC0-∞) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  AUC0-∞ of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Apparent terminal half-life (t1/2,λz) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  t1/2,λz (calculated from (ln 2)/λz being the apparent terminal rate constant) of GLPG0634 and its metabolite after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Metabolite over parent ratio of AUC0-24h (R) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  R (metabolite over parent ratio of AUC0-24h) after single and multiple dosing in subjects with renal impairment versus subjects with normal renal function
Accumulation ratio (Rac) | Between Day 1 at pre-dose up to 168 h after the last dose on Day 10 (Day 17)
  Rac (calculated as AUC0-24h Day 10/AUC0-24h Day 1) after dosing in subjects with renal impairment versus subjects with normal renal function
The number of subjects with adverse events | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 in subjects with renal impairment versus subjects with normal renal function in terms of adverse events (AEs)
The number of subjects with abnormal laboratory parameters | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 in subjects with renal impairment versus subjects with normal renal function in terms of abnormal laboratory parameters
The number of subjects with abnormal vital signs | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 in subjects with renal impairment versus subjects with normal renal function in terms of abnormal vital signs
The number of subjects with abnormal electrocardiogram (ECG) | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 in subjects with renal impairment versus subjects with normal renal function in terms of abnormal electrocardiogram (ECG)
The number of subjects with abnormal physical examination | From screening up to 10 days after last dose (Day 20)
  To evaluate the safety and tolerability of GLPG0634 in subjects with renal impairment versus subjects with normal renal function in terms of abnormal physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Pille Harrison, MD, Study Director — Galapagos NV
Locations (1):
- CRS Clinical Research Services Kiel GmbH, Kiel, Germany